CLINICAL TRIAL: NCT00332683
Title: Endotracheal Tube Cuff Pressure Protocol to Reduce Dysphagia Following Anterior Cervical Spine Surgery: A Prospective Randomized Pilot Study
Brief Title: Reducing Dysphagia Associated With Anterior Cervical Spine Surgery by Maintaining Low Endotracheal Tube Cuff Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R-06-225; 12338
Record Dates: First submitted 2006-05-31; First posted 2006-06-02 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Deglutition Disorders
Keywords: Dysphagia; spine surgery; cuff pressure
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Patients randomly assigned to this group will have no changes in the ETT during surgery
  Interventions: Procedure: Maintaining a normal pressure in the ETT cuff
- Treatment group (Experimental): Patients in this group will undergo same surgery as control group but with a monitoring and manipulation of ETT pressure
  Interventions: Procedure: Maintaining low (15mmHg) ETT cuff pressure

INTERVENTIONS:
Procedure: Maintaining low (15mmHg) ETT cuff pressure — Manipulation of the ETT cuff pressure to hold a lower pressure of 15 mmHg
  Arms: Treatment group
Procedure: Maintaining a normal pressure in the ETT cuff — No manipulation to maintain a low pressure of 15 mm Hg in the ETT cuff
  Arms: Control

SUMMARY:
Anterior cervical spine surgery (ACSS) is one of the most common procedures performed by spinal surgeons. It is associated with a 30-50% risk of developing swallowing difficulties (dysphagia). Although these difficulties usually improve within 6 months, for some it remains a significant and persistent problem.

We hypothesize that lowering the cuff pressure will lower the risk of injury to soft-tissues in the neck that are important to swallowing function. Our objective in this study is to demonstrate a lower occurrence of swallowing problems after anterior cervical spine surgery in patients with lower endotracheal tube cuff pressure during surgery.

Forty patients will be randomly assigned to a treatment group or control group. The treatment group will have the cuff pressure maintained at 15mmHg during the entire duration of the procedure. The control group will have the cuff pressure monitored without manipulation. After surgery soft-tissue swelling will be assessed on the five routine neck x-rays taken. In addition, 3 questionnaires completed before surgery and at each scheduled follow-up appointment will measure and track changes in swallowing over time and assess the impact of swallowing function on the patient's overall health. The results of this study may show that making a minor, inexpensive change during an operation may lower the risk of swallowing difficulties after a relatively common surgery.

DETAILED DESCRIPTION:
Post-operative dysphagia is a well-documented complication of anterior cervical spine surgery (ACSS) with an estimated risk of 30 - 50% that patients will experience some degree of post-operative swallowing dysfunction. While symptoms often subside within 6 months the impact of swallowing difficulties may be far reaching within the health-care system. Patients may be at risk of aspiration pneumonia and require swallowing assessments and modified diets. These measures necessitate a prolonged hospital stay. Patients may be prescribed anti-inflammatory medications and steroids which can inhibit bony fusion, which is an essential component of healing and ensuring spinal stability following ACSS.

The ultimate goal of this project is to determine the effect of minimizing ETT cuff pressure on the frequency of post-operative dysphagia following ACD. We believe that maintaining the ETT cuff pressure at 15mmHg will decrease the incidence of post-operative dysphagia - a direct benefit to the patients in the treatment group. Maintaining the ETT cuff pressure at 15mmHg would require no additional intra-operative equipment or modification to existing equipment. This intervention would not modify standard operative practice or pose additional risks to patients. As a result the cost-to-benefit ratio of this intervention may be substantially favourable to patients and the health care system.

ELIGIBILITY:
Inclusion Criteria:

* Between 21 and 65 years of age
* Must be competent to give consent
* Undergoing a first time anterior cervical discectomy (ACD) with instrumentation to remove pressure from the nerve roots caused by bone spurs or herniated disc material which is documented by a diagnostic procedure (CT and/or MRI)*.
* Ability and willingness to participate in routine follow-up at 6 weeks, 3 months and 6 months following surgery*.

Exclusion Criteria:

* Previous anterior neck surgery
* Anterior neck malignancy
* Tracheostomy.
* Previous treatment for dysphagia
* Pregnancy
* Women of childbearing potential who are not using an effective method of contraception.
* Medical comorbidities (e.g. significant renal or hepatic disease) which, in the investigator's opinion, may interfere with the patient's suitability and participation in the study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-06-06 (Actual); Primary Completion 2013-07-31 (Actual); Study Completion 2013-07-31 (Actual)

PRIMARY OUTCOMES:
Severity of dysphagia | pre-operatively and at 24hrs, 6wks, 3mons and 6mons following surgery

SECONDARY OUTCOMES:
Overall health score | pre-operatively and at 24hrs, 6wks, 3mons and 6mons following surgery
Percentage change in anterior cervical soft-tissue thickness on plain lateral radiographs | pre-operatively and at 24hrs, 6wks, 3mons and 6mons following surgery
Cost-effectiveness | 6mons after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Neil Duggal, M.D., M.Sc., Principal Investigator — Lawson Health Research Institute, London Health Sciences Center
Locations (1):
- London Health Sciences Center, University Campus, London, Ontario, Canada

REFERENCES:
- [Background] Apfelbaum RI, Kriskovich MD, Haller JR. On the incidence, cause, and prevention of recurrent laryngeal nerve palsies during anterior cervical spine surgery. Spine (Phila Pa 1976). 2000 Nov 15;25(22):2906-12. doi: 10.1097/00007632-200011150-00012. PMID 11074678
- [Background] Bazaz R, Lee MJ, Yoo JU. Incidence of dysphagia after anterior cervical spine surgery: a prospective study. Spine (Phila Pa 1976). 2002 Nov 15;27(22):2453-8. doi: 10.1097/00007632-200211150-00007. PMID 12435974
- [Background] Frempong-Boadu A, Houten JK, Osborn B, Opulencia J, Kells L, Guida DD, Le Roux PD. Swallowing and speech dysfunction in patients undergoing anterior cervical discectomy and fusion: a prospective, objective preoperative and postoperative assessment. J Spinal Disord Tech. 2002 Oct;15(5):362-8. doi: 10.1097/00024720-200210000-00004. PMID 12394659
- [Background] Ratnaraj J, Todorov A, McHugh T, Cheng MA, Lauryssen C. Effects of decreasing endotracheal tube cuff pressures during neck retraction for anterior cervical spine surgery. J Neurosurg. 2002 Sep;97(2 Suppl):176-9. doi: 10.3171/spi.2002.97.2.0176. PMID 12296675
- [Background] Riley LH 3rd, Skolasky RL, Albert TJ, Vaccaro AR, Heller JG. Dysphagia after anterior cervical decompression and fusion: prevalence and risk factors from a longitudinal cohort study. Spine (Phila Pa 1976). 2005 Nov 15;30(22):2564-9. doi: 10.1097/01.brs.0000186317.86379.02. PMID 16284596
- [Background] Smith-Hammond CA, New KC, Pietrobon R, Curtis DJ, Scharver CH, Turner DA. Prospective analysis of incidence and risk factors of dysphagia in spine surgery patients: comparison of anterior cervical, posterior cervical, and lumbar procedures. Spine (Phila Pa 1976). 2004 Jul 1;29(13):1441-6. doi: 10.1097/01.brs.0000129100.59913.ea. PMID 15223936
- [Background] Sperry RJ, Johnson JO, Apfelbaum RI. Endotracheal tube cuff pressure increases significantly during anterior cervical fusion with the Caspar instrumentation system. Anesth Analg. 1993 Jun;76(6):1318-21. doi: 10.1213/00000539-199376060-00023. PMID 8498671
- [Background] Tu HN, Saidi N, Leiutaud T, Bensaid S, Menival V, Duvaldestin P. Nitrous oxide increases endotracheal cuff pressure and the incidence of tracheal lesions in anesthetized patients. Anesth Analg. 1999 Jul;89(1):187-90. doi: 10.1097/00000539-199907000-00033. PMID 10389801
- [Background] Vanderveldt HS, Young MF. The evaluation of dysphagia after anterior cervical spine surgery: a case report. Dysphagia. 2003 Fall;18(4):301-4. doi: 10.1007/s00455-003-0012-z. PMID 14571336